CLINICAL TRIAL: NCT05347849
Title: A Two-part Phase 1, Single Ascending Dose Study to Evaluate the Safety, Tolerability and Pharmacokinetic Profile of Intranasal BPL-003 (5-Methoxy-N,N-dimethyltryptamine Benzoate) in Healthy Subjects
Brief Title: Single Ascending Dose Study With BPL-003 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beckley Psytech Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BPL-003-103
Record Dates: First submitted 2022-04-21; First posted 2022-04-26 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Pharmacokinetics in Healthy Adults

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part A only
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BPL-003 arm (Experimental)
  Interventions: Drug: BPL-003
- Placebo arm (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: BPL-003 — A single dose of BPL-003 will be administered intranasally
  Arms: BPL-003 arm
Other: Placebo — A single dose of placebo will be administered intranasally
  Arms: Placebo arm

SUMMARY:
The study will evaluate safety, tolerability and PK profile of BPL-003 in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* Medically healthy based on medical records and study specific assessments

Exclusion Criteria:

* Presence or history of severe adverse reaction to any drug or drug excipient

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2024-01-19 (Actual); Study Completion 2024-01-19 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with treatment emergent AEs (TEAES) | From screening through to the follow up visit, up to 65 days

SECONDARY OUTCOMES:
Peak plasma concentration (Cmax) | Day 1 (dosing day) and Day 2
Time to reach Cmax (tmax) | Day 1 (dosing day) and Day 2
Area under the plasma concentration- time curve | Day 1 (dosing day) and Day 2

CONTACTS AND LOCATIONS:
Overall Officials: VP & Head of Clinical Development, PhD, Study Director — Beckley Psytech Ltd
Locations (1):
- Hammersmith Medicines Research, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Due to the UK GDPR, individual participant data will not be shared publicly. Group data will be presented in publication after study completion

REFERENCES:
- [Derived] Rucker JJ, Roberts C, Seynaeve M, Young AH, Suttle B, Yamamoto T, Ermakova AO, Dunbar F, Wiegand F. Phase 1, placebo-controlled, single ascending dose trial to evaluate the safety, pharmacokinetics and effect on altered states of consciousness of intranasal BPL-003 (5-methoxy-N,N-dimethyltryptamine benzoate) in healthy participants. J Psychopharmacol. 2024 Aug;38(8):712-723. doi: 10.1177/02698811241246857. Epub 2024 Apr 14. PMID 38616411